CLINICAL TRIAL: NCT02998931
Title: Effects of Enteral Glutamine on Inflammatory Response, Immune System Function and Clinical Outcomes in Hospitalized Patients With Enteral Feeding in Intensive Care Unit
Brief Title: Trial of Enteral Glutamine on Clinical Outcomes in Critically Ill Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate Professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1395/670
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Critical Illness; Enteral Nutrition; Multiple Organ Failure; Infection Complication; Inflammation
Keywords: Glutamin; Enteral Nutrition; Intensive Care Unit; Critical Care Outcomes; inflammatory; Immune System
MeSH Terms: conditions — Critical Illness; Multiple Organ Failure; Inflammation | interventions — glutamin-(asparagin-)ase; Glutamine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamin (Experimental): Intervention patients will be received enteral formula and glutamine 0.3 g/kg/day given via nasogastric tube as boluses q 4hrs.
  Interventions: Drug: Glutamin
- maltodextrin (Placebo Comparator): Control patients will be received enteral formula and maltodextrin mixed in with water and given via nasogastric tube as boluses q 4hrs.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Drug: Glutamin — Enteral Glutamine 0.3g/kg/day powdered glutamine to be mixed in with water and given via nasogastric tube q4 hrs
  Other Names: L-glutamine
  Arms: Glutamin
Other: Maltodextrin — Maltodextrin mixed with water given via NG tube Q 4 hours
  Arms: maltodextrin

SUMMARY:
Glutamine supplementation has beneficial effects on morbidity and mortality in critically ill patients, possibly in part through an attenuation of the proinflammatory cytokine response and a Immune function. In this trial intensive care unit patients with enteral feeding will receive either enteral glutamine or maltodextrin as placebo for 28 days.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in general intensive care unit (ICU) in Tehran, Iran. After a full review of the inclusion and exclusion criteria and explanation of the risks and benefits of the study, written consent form will be completed. The participants are 200 eligible hospitalized patients with enteral feeding in ICU, aged ≥ 18 years. Intervention patients will be received 0.3 g/kg/day of glutamine along with enteral formula for 28 days and control patients will be received maltodextrin along with enteral formula for 28 days. Patients will be evaluated for occurrence of new infection, organ failure, duration of stay in ICU, 28 days and 6 months mortality and inflammatory and immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) admitted to ICU
* Start of study intervention within 48 hours after ICU admission
* Expected to require enteral nutrition for at least 72 hours aiming for full enteral nutrition and receive at least 80 percent of enteral formula during the first 48 hour
* Written informed consent of patient or written informed consent of legal representative

Exclusion Criteria:

* Enrollment in a related ICU interventional study
* Requiring other specific enteral nutrition for medical reason
* Death or Discharge before 5th day
* Having any contra-indication to receive enteral nutrition
* Pregnant patients or lactating with the intent to breastfeed
* Requiring other specific enteral nutrition for medical reason
* BMI <18 or > 40.0 kg/m2
* Have life expectancy of <6 mo
* Patients who are moribond
* Liver cirrhosis- Child's class C liver disease
* Have seizure disorder requiring anticonvulsant
* History of allergy or intolerance to the study product components
* Receiving glutamine during two weeks before start study product
* Have other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of infection | Day 28
  Incidence of infections

SECONDARY OUTCOMES:
Serum Inflammatory Markers | baseline, Day 5, Day 10
  Inflammatory factors
Serum Immunity Markers | baseline, Day 5, Day 10
Length of stay in ICU | Day 28
28-day Mortality | Day 28
  Day 28
6-month mortality | month 6
  month 6

OTHER OUTCOMES:
Serum Glutamin | baseline, Day 5, Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, MD, PhD, Study Chair — Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (2):
- Iran (2):
  - Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran
  - Shohada Tajrish Hospital, Tehran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Zanten AR, Sztark F, Kaisers UX, Zielmann S, Felbinger TW, Sablotzki AR, De Waele JJ, Timsit JF, Honing ML, Keh D, Vincent JL, Zazzo JF, Fijn HB, Petit L, Preiser JC, van Horssen PJ, Hofman Z. High-protein enteral nutrition enriched with immune-modulating nutrients vs standard high-protein enteral nutrition and nosocomial infections in the ICU: a randomized clinical trial. JAMA. 2014 Aug 6;312(5):514-24. doi: 10.1001/jama.2014.7698. PMID 25096691
- [Background] Heyland D, Muscedere J, Wischmeyer PE, Cook D, Jones G, Albert M, Elke G, Berger MM, Day AG; Canadian Critical Care Trials Group. A randomized trial of glutamine and antioxidants in critically ill patients. N Engl J Med. 2013 Apr 18;368(16):1489-97. doi: 10.1056/NEJMoa1212722. PMID 23594003
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Kreymann KG, Berger MM, Deutz NE, Hiesmayr M, Jolliet P, Kazandjiev G, Nitenberg G, van den Berghe G, Wernerman J; DGEM (German Society for Nutritional Medicine); Ebner C, Hartl W, Heymann C, Spies C; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Intensive care. Clin Nutr. 2006 Apr;25(2):210-23. doi: 10.1016/j.clnu.2006.01.021. Epub 2006 May 11. PMID 16697087
- [Background] McQuiggan M, Kozar R, Sailors RM, Ahn C, McKinley B, Moore F. Enteral glutamine during active shock resuscitation is safe and enhances tolerance of enteral feeding. JPEN J Parenter Enteral Nutr. 2008 Jan-Feb;32(1):28-35. doi: 10.1177/014860710803200128. PMID 18165444
- [Background] Hall JC, Dobb G, Hall J, de Sousa R, Brennan L, McCauley R. A prospective randomized trial of enteral glutamine in critical illness. Intensive Care Med. 2003 Oct;29(10):1710-6. doi: 10.1007/s00134-003-1937-2. Epub 2003 Aug 16. PMID 12923621